CLINICAL TRIAL: NCT00417820
Title: A Multicenter, Double-Blind, Placebo Controlled Exploratory Study to Evaluate the Safety, Tolerability and Pharmacodynamics of a Single Administration of BCT194 in Healthy Volunteers and Multiple Administrations in Patients With Psoriasis.
Brief Title: Study of the Safety, Tolerability and Efficacy of BCT194 in Healthy Volunteers and Patients With Psoriasis.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBCT194A2101
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Last update posted 2007-11-29 (Estimated); Status verified 2007-11

CONDITIONS: Psoriasis
Keywords: Safety, tolerability, pharmacodynamics, single administration, BCT194, healthy volunteers, psoriasis
MeSH Terms: conditions — Psoriasis

INTERVENTIONS:
Drug: BCT194

SUMMARY:
The purpose of this study is to assess the local tolerability of a single topical administration of BCT194 in healthy volunteers and, potentially, to evaluate the safety, tolerability, and efficacy of a multiple topical administrations in patients with psoriasis.

ELIGIBILITY:
Inclusion Criteria:

All participants:

* Healthy male and female (of non-childbearing potential) subjects age 18 to 45 years of age included, and in good health as determined by past medical history Postmenopausal women must have had no regular menstrual bleeding for at least 1 year prior to inclusion or female subjects must have been surgically sterilized at least 6 months prior to screening supported by clinical documentation.

Male subjects must be using a double-barrier local contraception.

* Body weight must be between 50 and 100kg (inclusive) to participate in this study
* Able to communicate well with the investigator, to understand and comply with the requirements of the study. Understand and sign the written informed consent.

Psoriasis patients:

* Diagnosis of stable plaque psoriasis with or without arthritis for at least 6 months prior to screening.
* Absence of clinically relevant abnormalities for screening laboratory test results of hematological (hemoglobin, white blood cells, neutrophils, platelets), renal (serum creatinine) and hepatic (aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, gammaglutamyltransferase,bilirubin) parameters.
* Willingness to avoid sunbeds or unusual sun exposure during the study period.

Exclusion Criteria:

All participants:

* Use of any prescription drugs within 4 weeks prior dosing, or over-the-counter medication (vitamins, herbal supplements, dietary supplements) within 2 weeks prior to dosing. Paracetamol is acceptable,
* Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulations, and for any other limitation of participation based on local regulations.
* Donation or loss of 400 ml or more of blood within 8 weeks prior to first dosing, or longer if required by local regulation.
* Significant illness within two weeks prior to dosing.
* A past personal or close family medical history of clinically significant cardiac abnormalities
* History of:

  * Acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease)
  * Clinically significant drug allergy or history of atopic allergy (asthma, urticaria, eczematous dermatitis)
  * Known hypersensitivity or severe adverse event to darifenacin or similar drugs
  * Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or which may jeopardize participation in the study
  * Immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result
  * Positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.
  * Drug or alcohol abuse within the 6 months prior to dosing.
* History of abnormal skin reactivity to UV light. Unusual exposure to UV light in the previous 3 weeks prior to study start, including tanning, sunbeds etc.

Psoriasis patients:

* Currently have any of the nonplaque forms of psoriasis: erythrodermic, guttate, or pustular.
* Currently have drug-induced psoriasis (new onset or exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium).
* Used any investigational drug within the previous 4 weeks.
* Recent previous treatment with anti-TNF-α therapy (or other biological therapy),immunosuppressive agents such as cyclosporine, mycophenolate, pimecrolimus, or tacrolimus.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2006-11; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Safety & tolerability
Efficacy as assessed by plaque Psoriasis Area and Severity Index (PASI) scoring at 4 weeks

SECONDARY OUTCOMES:
Potential of absorption of topical BCT194 into the systemic circulation and to determine skin exposure
Cellular changes in psoriasis skin by immunohistology at day 8
Changes in HSP-27 and phospho (p) HSP-27 in protein lysates of skin biopsies at Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigator site
Locations (1):
- Novartis Investigative Site, Vienna, Austria